CLINICAL TRIAL: NCT06194370
Title: The Application of BOPPPS（Bridge-in,Objective,Pre-assessment,Participatory Learning,Post-assessment,Summary） Model in the Ward Rounds of Nurses' Standardized Training
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: First Affiliated Hospital of Chongqing Medical University (Other)
Responsible Party: Principal Investigator, Ying Shen, Study Director, First Affiliated Hospital of Chongqing Medical University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: K2023-191
Record Dates: First submitted 2023-12-14; First posted 2024-01-08 (Actual); Last update posted 2024-01-08 (Actual); Status verified 2024-01

CONDITIONS: Standardized Training

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BOPPPS Teaching Model Group (Experimental): BOPPPS: Bridge-in,Objective,Pre-assessment,Participatory learning,Post-assessment,Summary
  Interventions: Other: Training by BOPPPS Teaching Model
- Regular Teaching Group (Placebo Comparator)
  Interventions: Other: Training Regularly

INTERVENTIONS:
Other: Training by BOPPPS Teaching Model — Training by BOPPPS Teaching Model
  Arms: BOPPPS Teaching Model Group
Other: Training Regularly — Training Regularly
  Arms: Regular Teaching Group

SUMMARY:
Nursing standardization training students in a top-three hospital in Chongqing from July 2017 to June 2022 were selected as the research objects, excluding nursing students who participated in online courses during the epidemic period. The BOPPPS(Bridge-in,Objective,Pre-assessment,Participatory learning,Post-assessment,Summary) teaching model was applied to the standardized training of nurses and compared with the conventional teaching methods to evaluate the effect of improving the theoretical knowledge, professional skills and comprehensive ability of nursing students.

ELIGIBILITY:
Inclusion Criteria:

* Nursing standardization training students in a top-three hospital in Chongqing

Exclusion Criteria:

* Nursing students who participated in online courses during the epidemic period

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2024-01 (Estimated)

PRIMARY OUTCOMES:
Comprehensive ability evaluation | 1 month
  Using 5-point Likert scale to evaluated comprehensive ability.A higher score indicated a higher comprehensive competence

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality, China